CLINICAL TRIAL: NCT07264023
Title: A Prospective, Observational, Multicenter Longitudinal Cohort Study on the Correlation Between Nutritional Status and Quality of Life in Children With Neuro-oncological Tumors During the Peri-radiotherapy Period.
Brief Title: Correlation Between Nutritional Status of Childhood Neurological Tumors and Quality of Life
Status: Not yet recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2025-582
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Nutritional Status; Quality of Life; Children; Brain Tumor, Primary
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Maintaining good nutritional status during treatment for children with cancer is crucial for many outcomes, such as overall survival rate, tolerance to treatment, susceptibility to infection, and quality of life. Neurotumors in children account for the highest proportion among solid tumors in children. Previous studies have clearly shown that neurotumors in children have different nutritional characteristics from hematological tumors and other solid tumors in children. Our retrospective data found that there was a significant correlation between the BMI Z values of children with neurotumors before and during radiotherapy and the frequency of adverse events. The occurrence of adverse events has a negative impact on the quality of life of child patients. Therefore, we plan to conduct a prospective, observational, multi-center longitudinal cohort study to evaluate the dynamic changes in nutritional status during the peri-radiotherapy period, explore the correlation between nutritional status and quality of life in children with neurotumors before and after radiotherapy, and establish a nutritional management plan and nutritional risk early warning model suitable for Chinese children with neurotumors.

ELIGIBILITY:
Inclusion Criteria:

* The patient and the legal guardian have agreed to sign the informed consent form;
* Age ≥ 5 years old and ≤ 18 years old;
* The pathological or clinical diagnosis is a neurological tumor;
* Patient has indications for radiotherapy;
* The expected survival time is over 6 months.

Exclusion Criteria:

* Accompanied by other serious complications;
* The researcher judged that it was not suitable to participate in this study.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children with neuro-oncological tumors
Sampling Method: Non-Probability Sample
Enrollment: 93 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
life quality | Before radiotherapy, at the end of radiotherapy, one month after radiotherapy, three months after radiotherapy, six months after radiotherapy
  The PedsQL Brain Tumor Module and the PedsQL4.0 Generic Core Scale for Children were used to assess the quality of life of the subjects. The assessment data were collected, including the children's self-assessment module and the parent proxy assessment module, covering dimensions such as physical function, emotional function, social function, and school function.
nutritional status | Before radiotherapy, at the end of radiotherapy, one month after radiotherapy, three months after radiotherapy, and six months after radiotherapy